CLINICAL TRIAL: NCT06425627
Title: Spinal Versus General Anesthesia on Postoperative Pulmonary Complications in Elderly Patients With Delayed Operation of Hip Fracture
Brief Title: Spinal Versus General Anesthesia on Postoperative Pulmonary Complications
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Tianzhu Liu, M.D., Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TongjiHospital102114
Record Dates: First submitted 2024-05-09; First posted 2024-05-22 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Complication; Anesthesia; Hip Fractures
Keywords: Hip fracture; delayed surgery; pulmonary complication; spinal anesthesia; general anesthesia
MeSH Terms: conditions — Hip Fractures | interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- spinal anesthesia (Experimental): Patients underwent real-time ultrasound guided spinal anesthesia. The maximum attempts of skin piercings are 3, and the total redirections of each skin piercings should not exceed 6 times. General anesthesia was considered if three skin piercings were unsuccessful.
  Interventions: Procedure: spinal anesthesia
- general anesthesia (Experimental): Rapid sequential induction was performed with sufentanil 0.5 ug /kg, etomidate 0.3 mg /kg, cisatracurium 0.15 mg /kg, and then laryngeal mask was applyed. Parameter settings: tidal volume: 6-10 mL/kg, 1.5 ~ 2.0% sevoflurane inhalation, remifentanil 0.1 ~ 0.2 ug/ kg.min-1. Mechanical driving pressure was applyed by PEEP titration method.
  Interventions: Procedure: general anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — An intrathecal anesthetic technique.
  Other Names: lumbar anesthesia
  Arms: spinal anesthesia
Procedure: general anesthesia — An intravenous (combined with inhalation) anesthetic technique.
  Arms: general anesthesia

SUMMARY:
The objective of this study was to investigate the difference in postoperative pulmonary complications (PPCs) between spinal anesthesia and general anesthesia in patients undergoing delayed hip surgery.

DETAILED DESCRIPTION:
In this study, the difference of 30 min arterial partial pressure of oxygen after operation was used as the main outcome index. By means of pulmonary ultrasound, pulmonary function monitoring and other physical and biochemical examinations, the difference of postoperative pulmonary complications between spinal anesthesia and general anesthesia in patients with delayed operation of hip fracture longer than 48 hours was compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 65 years old
* ASA Class I ~ III
* Surgical repair of femoral neck, intertrochanteric or subtrochanteric fractures
* The time from diagnosis to surgery is more than 48 hours

Exclusion Criteria:

* Unable to walk about 3 meters or across a room without assistance before the fracture
* Emergency surgery
* Congestive heart failure, asthma, anemia (Hb < 90 g/L), hypoalbuminemia (ALB < 35g/L)
* Abnormal coagulation function
* Severe aortic stenosis
* Injection site infection or increased intracranial pressure
* Patients have participated in previous trials or have been determined by a surgeon or anesthesiologist to be unsuitable for randomization
* The written informed consent of the patient or his/her representative cannot be obtained

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Arterial partial pressure of oxygen, PaO2 | 30 minutes after surgery
  PaO2 was measured by arterial blood gas analysis

SECONDARY OUTCOMES:
Arterial partial pressure of oxygen, PaO2 | 30 minutes before surgery
  PaO2 was measured by arterial blood gas analysis
Forced vital capacity, FVC | 30 minutes before surgery; 30 minutes after surgery; 24 hours after surgery
  FVC was measured by Spirometer (SP70B)
Forced expiratory volume in 1 second, FEV1 | 30 minutes before surgery; 30 minutes after surgery; 24 hours after surgery
  FEV1 was measured by Spirometer (SP70B)
Peak expiratory flow, PEF | 30 minutes before surgery; 30 minutes after surgery; 24 hours after surgery
  PEF was measured by Spirometer (SP70B)
PEF 25, 75, and 25-75 | 30 minutes before surgery; 30 minutes after surgery; 24 hours after surgery
  PEF 25, 75, and 25-75 were measured by Spirometer (SP70B)
Lung Ultrasound Score (LUS) | 30 minutes before surgery, 30 minutes after surgery, 24 hours after surgery
  Bedside measurements using portable ultrasound
Postoperative pulmonary complications | up to one month
  Pulmonary complications (PPCs) include: (1) Evidence of pneumonia, pneumothorax, atelectasis and pleural effusion indicated by postoperative pulmonary ultrasound, chest film or chest CT; ② After surgery, the patient developed bronchospasm, ARDS, O2 requirement (nasal catheter or mask), non-invasive ventilation requirement, or unplanned endotracheal intubation/mechanical ventilation for more than 1 day; ③ The increase of inflammatory biochemical indexes 24 h after surgery suggested systemic inflammatory response (blood routine, C-reactive protein CRP, procalcitonin PCT and IL-6, IL-1β, TNF-α).
Hip mobility (Harris hip score, HHS) | up to one month
  The Harris scale was used to score. Range:0-100. A total Harris hip score below 70 points was considered a poor result, 70 to 80 fair, 80 to 90 good, and 90 to 100 excellent.

OTHER OUTCOMES:
Adverse outcomes | up to one month
  Documented side effects associated with the intervention by an unwitting third party

CONTACTS AND LOCATIONS:
Overall Officials: Tianzhu Liu, M.D., Principal Investigator — Tongji Hospital
Locations (1):
- Tianzhu Liu, Wuhan, Hubei, China